CLINICAL TRIAL: NCT02590822
Title: Diabetes Interventional Assessment of Slimming or Training to Lessen Inconspicuous Cardiovascular Dysfunction. The Diastolic Study
Brief Title: Diabetes Interventional Assessment of Slimming or Training to Lessen Inconspicuous Cardiovascular Dysfunction
Acronym: Diastolic
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Leicester (Other)
Collaborators: University Hospitals, Leicester (Other); National Institute for Health Research, United Kingdom (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0498; 182089 (Other: NIHR Clinical Research Network)
Record Dates: First submitted 2015-10-19; First posted 2015-10-29 (Estimated); Last update posted 2024-01-05 (Actual); Status verified 2024-01

CONDITIONS: Diabetes
Keywords: Diabetes; T2DM; young adults; heart; weight loss; MRI; exercise; diastolic function
MeSH Terms: conditions — Diabetes Mellitus; Weight Loss; Motor Activity | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Standard Care (No Intervention): The Standard Care group will be contacted weekly (where possible) to reinforce cognitive behavioural adaptations and encourage compliance to diet and exercise. They will be provided with standard lifestyle advice according to NICE guidance.
- Total Dietary Replacement (Experimental): Group receives a total meal replacement diet from Cambridge Weight Plan containing 810 kcal/day (40% protein, 50% carbohydrate, 10% fat). The diet will be stopped, and a maintenance diet re-introduced once 50% excess body weight has been lost, or by 12 weeks, whichever comes first.
  The TDR will be undertaken alongside health behaviour coaching and relapse prevention contact & current medications will need to be adjusted initially and throughout the study.
  Interventions: Dietary Supplement: Cambridge Weight Plan
- Supervised Exercise (Experimental): The exercise group will attend thrice weekly 60minute supervised exercise sessions at the Leicester-Loughborough Diet, Lifestyle and Physical Activity (LLP) BRU or at the Leicester Diabetes Centre. An initial assessment of cardiorespiratory fitness will be performed (VO2 max) to allow design of a tailored exercise programme.
  Current medication will need to be adjusted initially and throughout the study.
  Interventions: Other: Supervised Exercise Sessions

INTERVENTIONS:
Dietary Supplement: Cambridge Weight Plan — Group receives a total meal replacement diet from Cambridge Weight Plan containing 810 kcal/day (40% protein, 50% carbohydrate, 10% fat). As 3 or 4 mini-meals daily in flavoured formula food packets made up with water, milk or non-dairy alternative; or as snack bars based on preference. Supplemented with up to three portions of non-starchy vegetables and 2 litres of water, or other non-calorific drinks, per day. Participants to abstain from alcohol for study duration. The diet will be stopped, and a maintenance diet re-introduced once 50% excess body weight has been lost, or by 12 weeks, whichever comes first.
  The TDR will be undertaken alongside health behaviour coaching and relapse prevention through weekly, where possible, contact (telephone or face-to-face) with a qualified dietician or equivalent.
  Due to the potential risk of hypoglycaemia and symptomatic hypotension; medication at enrolment will need to be adjusted initially and throughout the study.
  Arms: Total Dietary Replacement
Other: Supervised Exercise Sessions — The exercise group will attend supervised exercise sessions at the Leicester-Loughborough Diet, Lifestyle and Physical Activity (LLP) BRU or at the Leicester Diabetes Centre. The exercise program will typically consist of a thrice weekly, 60 minute session of moderate intensity aerobic exercise, in line with prevailing guidelines. An initial assessment of cardiorespiratory fitness will be performed, and exercise intensity titrated to aim for a workload of approximately 60% of the patient's VO2 max.
  Due to the potential risk of hypoglycaemia and symptomatic hypotension; medication at enrolment will need to be adjusted initially and throughout the study.
  Other Names: Physical Activity
  Arms: Supervised Exercise

SUMMARY:
There is an epidemic of type 2 diabetes in younger adults. These patients are at very high lifetime risk of heart-related complications. Subtle heart abnormalities can be present even at a young age in these patients and may predispose them to heart failure and ultimately premature death. There is emerging evidence that type 2 diabetes can be reversed with weight loss. We propose that weight loss can also reverse the fatty changes seen in the liver and heart in these patients, and in turn lead to improved heart function.

This project aims to identify how type 2 diabetes causes changes in the heart in young people with type 2 diabetes by performing detailed scans and other tests of the heart's structure and function. In addition we will attempt to see if the heart's pumping function can be improved, either by a weight loss program with a special low calorie diet, or by a structured program of exercise. This will be compared with the usual standard diabetes care.

As well as looking to see if the heart's function can be improved with the intervention, we also aim to identify what the mechanism of any improvement would be. We suspect that changes in the amount of fat within the liver and the heart may be responsible, and will measure these at the beginning, end and in some patients halfway through the study to explore possible mechanisms amongst other clinical variables (e.g. HbA1c)

DETAILED DESCRIPTION:
This is a single centre study, which will comprise of a cross-sectional analysis of the baseline data of a 3-arm 12 week Prospective, Randomised, Open label, Blinded End point (PROBE) trial of TDR and an exercise programme compared with standard care. Clinical follow-up will take place at 6-12 months.

The trial has two primary objectives:

1) Identify the determinants of diastolic dysfunction, assessed by MRI, in younger adults with T2DM through multivariate analysis of baseline dataset (cross-sectional study analysis) 2) Determine if diastolic dysfunction (classified by diastolic strain rate) can be reversed by either TDR or an exercise programme (PROBE trial)

Secondary objectives include:

1. Determine the reference range for diastolic strain rate in healthy adults
2. Determine the optimum field strength for the assessment of PEDSR

   * Sample size:

   Cross-sectional Analysis: A sample size of 100 T2DM participants will have approximately 80% power to test up to 10 variables in a multivariate regression analysis, with an estimated combined R2 of 15%, for the identification of determinants of diastolic stain rate.

   - PROBE Trial:

   All participants from Phase I who agree to take part in Phase II will be randomized. The Investigators expect, based on experience from previous studies, an attrition rate of up to 10% following the first data collection session. Therefore, approximately 90 participants are expected to be randomized to the three arms (approximately 30/group). The power calculation is based on the Investigators pilot MRC study. The T2DM patients had diastolic strain rate of 1.5s-1 with standard deviation of 0.2 s-1. Based on this, 30 patients per group will have 80% power to detect a between group difference in peak early diastolic strain rate (PEDSR) of 0.2s-1 assuming alpha=0.025 (to allow for two primary comparisons, i.e. TDR vs standard care and exercise vs standard care) and a maximum 30% drop-out. Such an improvement would result in a strain rate (1.7 s-1) similar to that seen in the obese controls (1.8 s-1) but still lower than the lean controls (2.0 s-1).
   * Randomization:

   Randomization will be stratified by sex, given different left ventricular remodeling processes in males and females, and by baseline glucose lowering therapy (any GLP-1, DPP-IV or SGLT-2 vs none of these). The statistician undertaking the final analysis will be blinded to the treatment groups.

   - Healthy controls:

   Twenty healthy controls will be recruited and undertake all baseline measures only. This population will serve to confirm normal ranges on the relevant scanners and will inform the cross-sectional analysis of baseline data and provide a comparator group for the study endpoints i.e. determine if the interventions have caused reversion to normal diastolic function in the T2DM population.

   - Test Re-Test MRI sub-study:

   An optional sub-study examining test-retest reproducibility of MRS at 1.5 and 3T will be performed on selected participants willing to undergo a second scan. Details of this sub-study are provided below. As outlined above our preferred field strength for the assessment of PEDSR is 1.5T. However, due to higher signal to noise of 3T imaging, MRS for myocardial triglyceride may be better at 3T but there have been no direct comparisons.

   Participants enrolled for the main study will be asked if they would be willing to take part in the reproducibility sub-study, until ten participants have been recruited. These participants will then undertake an additional 20 minute scan on the same on the 3T platform to assess myocardial triglyceride and PEDSR. The 3T scan will consist of localisers, cine long axis 4 chamber, 3 chamber and short axis at mid for calculation of myocardial strain rates as previously described, followed by single voxel H+ MRS of the interventricular septum to allow calculation of myocardial triglyceride content. No contrast will be administered during this examination.

   - Statistical Analysis:

   Cross-sectional Analysis:

   The aim of these analyses is to identify determinants of diastolic dysfunction in individuals with T2DM. Outcome and potential explanatory variables will be summarized using mean (standard deviation) for normally distributed continuous variables, median (interquartile range) for non-normally distributed continuous variables, and count (percentage) for categorical variables. We anticipate including the following potential explanatory variables: duration of diabetes, age, sex, myocardial and liver triglyceride content, myocardial perfusion reserve, blood pressure, HBA1c, blood pressure and myocardial extracellular volume. Univariate linear regression models will then be fitted with diastolic strain rate as the outcome, and each of the explanatory variables under consideration as the covariate in turn to identify factors associated with diastolic strain rate. Variables that have a significant univariate association with diastolic strain rate will be entered into a multivariate regression analysis to determine independent associations with diastolic strain rate. Redundant variables will be removed in a stepwise manner, based on a significance level of 0.05.

   - PROBE trial/Phase II:

   The aim of these analyses is to compare the primary outcome (diastolic strain rate) at 12 weeks between the TDR and standard care arms, and between the exercise and standard care arms. The primary analysis will be a per protocol analysis as this is a proof of principle study where we are primarily interested in the size of the treatment effect, rather than the practicability of the intervention. A CONSORT diagram will be produced. At baseline and each follow-up, outcome and descriptive variables will be summarized by arm using mean (standard deviation) for normally distributed continuous variables, median (interquartile range) for non-normally distributed continuous variables, and count (percentage) for categorical variables. Each intervention will be compared with the control group (i.e. TDR v standard care and Exercise v standard care) using linear regression to allow missing outcome data to be imputed using multiple imputation methods. If necessary, the outcome variable will be appropriately transformed so that the assumptions of the linear regression model are held.

   - Healthy controls:

   The aim of these analyses is to quantify the diastolic strain rate of healthy individuals as this is currently unknown. These analyses will provide context in which to interpret the results of the PROBE trial, and are not powered for a formal comparison between the T2DM patients and healthy controls as they are considered to be exploratory. A baseline summary of the outcome and descriptive variables used in the PROBE trial will be produced using mean (standard deviation) for normally distributed continuous variables, median (interquartile range) for non-normally distributed continuous variables, and count (percentage) for categorical variables.

   Should any unexpected and significant findings occur as a result of these tests, they will be communicated to the patients GP. This will be stated in the consent form for the healthy controls.

   - Test re-test:

   The aim of these analyses is determine whether diastolic strain rate measured on a 3T scanner (gold standard) is comparable with that measured on a 1.5T scanner. Descriptive characteristics of those participating in the test-retest sub-study will be summarized. Diastolic strain rate will be summarized using mean (standard deviation) or median (interquartile range), as appropriate, by scanner. Bland-Altman Limits of Agreement will be produced.

   The formal end of the study will occur following the final 12 week assessment of the final patient recruited

   We will conduct two further follow-up visits to assess maintenance at 6 and 12 months (or at study end). We will collect data for weight, blood pressure, lipid profile and glycaemic control. Patients will be asked to consent to the investigators accessing long-term follow-up (10 years) through review of clinical records and Hospital Episode statistics through flagging with the Health and Social Care Information Centre.
   * Study interventions:

   Recruited participants will be randomised to one of three groups for the PROBE study; 1. Standard of care as per NICE guidance plus lifestyle advice or 2. Total Dietary Replacement (TDR) or 3. Supervised exercise training.
   * Participant Compliance:

   TDR Group Participant Compliance:

   Previous studies with LED/VLED with TDR have indicated that compliance is between 70-80%. The patients in both the TDR and exercise groups will have regular contact with investigators to encourage compliance and offer support. The standard care group will also receive weekly telephone calls to encourage compliance to suggested lifestyle changes. Participants will be offered £50 compensation for completing each of the three assessments, which will take approximately 3-4 hours. However, those patients in the TDR arm that do not achieve a loss of >4% body weight at week 1 and 10% at week four will be considered non-compliant and excluded from the study.

   Exercise Group Participant Compliance:

   Compliance will be assessed by attendance at the supervised sessions. Participants in the exercise arm who attend less than two thirds of the supervised sessions in the first 4 weeks will be excluded (PI discretion will be applied to this determination where necessary).

   - Alterations to medication regime:

   Due to the potential risk of hypoglycaemia and symptomatic hypotension; medication at enrolment will need to be adjusted initially and throughout the study for both the TDR and the exercise training groups.

   Participants randomised to the TDR group:Will be asked to discontinue with all glucose lowering therapies before the baseline study, as previously advised for a recently published study with similar intervention (of 8 weeks). Metformin and Sulphonylureas are to be discontinued 72hours prior to initiation of TDR. DPP IV inhibitors 2, GLP-1 therapies and SGLT2s will be discontinued 2 weeks prior to the initiation of the TDR. Antihypertensive drugs will be stopped on the day the TDR is commenced. This is a safety measure because blood pressure is likely to fall substantially (mean drop in SBP ~ 20mmHG) on the diet. Medication will be adjusted DiRECT study protocol (see supplementary material) however, individual clinical decisions may be necessary for a patient's best interest and therefore any alterations to medication are ultimately made at the discretion of the study clinician(s). Blood pressure will be monitored throughout the study at the clinical review sessions as per the DiRECT protocol. Treatments for other conditions and primary prevention of cardiovascular disease (e.g. statins) will be continued. This will be discussed in detail and decided upon at the level of the individual, at the initial consultation. Furthermore, their medical history will be taken and any participant with a history of constipation other bowl related problems will be prescribed a fibre supplement i.e. fybogel to help to prevent its occurrence. We will ask participants to continue with their habitual levels of physical activity throughout the course of the study.

   Participants who achieve a 50% reduction in excess body mass before completion of the 12-week programme will revert to a maintenance diet and will complete the assessments at 12 weeks.

   Participants randomised to exercise training: Will have their medication reviewed by the study clinician. Those with a HbA1c ≤ 8% who are currently taking a sulphonylurea will initially have the dose reduced by 50% 72hours prior to the first exercise session. Their regimes will be continued to be down titrated starting with the sulphonylurea and then moving, where applicable, onto their current SGLT or DPP-IV or GLP-1 therapies according to glycaemic control. The latter therapies will be titrated down last given their relative low risk of hypoglycaemic events. For those participants with a HbA1c ≤ 8% who are not taking a sulphonylurea the study clinician will down titrate glucose-lowering therapy on an individual basis, taking into account the class and combination of therapies prescribed. All other medication will be maintained unless the study clinician deems alterations are necessary for a patient's best interest. Any alterations will be recorded in the CRF and statistically adjusted for in the analysis.

   - Psychological support:

   This support will be provided in the form of a health coaching approach with the inclusion of relapse prevention strategies. This model of working is based upon a patient centered approach that employs principles from health psychology and behavioral medicine, and the skills and attitude from health coaching and motivational interviewing. The aim is to focus upon the participants own intrinsic motivators, explore barriers and encourage the development of personally determined solutions. The initial clinical consultation will allow a review of the participant's gains from engaging in the TDR or training programme and potential barriers that may arise and individualise solutions. This will be recorded for the participant to take away and will form the basis of the telephone/face to face follow up and group support. There is a convergence of evidence from multiple sources that these approaches beneficially impact behavioural change.

   - Participant clinical review:

   All participants will have an initial clinical review post-randomisation at the time of their health coaching. In order to ensure the continued safety of each participant following the discontinuation and/or reduction in mediation regime they will be invited for a basic clinical review once a week for the first four weeks and fortnightly thereafter. They will attend six reviews after randomisation in total (weeks 1,2,4,6,8, and 12), as well as receiving a telephone consultation at weeks 3 and 10. At these clinical reviews their blood pressure, fasting glucose and weight will be measured. This is to inform; a) any additional alterations to medication that need to be made and b) compliance to TDR (if in that group). In addition, all participants will have access to telephone support from the diabetes team in the case of any symptoms or concerns over glycaemic control. The reviews will be performed by a qualified nurse, under the supervision of a study clinician specialised in diabetic medicine at the Leicester Diabetes Centre. Any changes to medication made at these visits will be communicated to the patients GP by letter.

   At the end of the 12 week intervention all participants' medication will be reviewed again and any medication re-introduced will be tailored to the individual based on previous and current HbA1c and blood pressures. This review will be undertaken by an experienced study clinician(s) and the outcome communicated to the patient's usual physician and GP.

   - Blood glucose monitoring:

   Each participant will be provided with the provisions to enable multiple daily finger-stick testing which they can record in a standardized blood glucose diary that will be provided. This will allow us to capture any hypoglycaemic events (as defined below) and adjust medication accordingly if required. We will additionally be able to capture any hyperglycaemia which can again be addressed by alterations to medication and review of compliance to intervention. In addition, glycaemic control will be monitored at clinical review sessions with fasting glucose and HbA1c levels.

   - Recruitment strategies:

   The recruitment phase will commence as soon as ethical, research governance and regulatory approval has been granted. Potential participants will be identified and approached to participate in this study from a number different settings as outlined below. It is envisaged that those participating in phase I will enter into phase II of the study and therefore these strategies are applicable to both phases.

   We have extensive links across primary care that we will draw upon for this study. We will target specialist's diabetes outpatient clinics located in the community (for example Hinckley, Melton Mowbray and Oakham), the intermediate Care Division (ICD) for diabetes and secondary care.We have good links with the Leicester Royal Infirmary bariatric surgery service where a large cohort of eligible people exists on the referral list for surgery.Potentially eligible patients who have previously participated in other research studies at the LDC and have indicated a willingness to take part in additional studies will also receive a postal invite. We hold a volunteer database with the contact information and basic data of people who have expressed an interest in participating in more research further, we have a list of young adults with T2DM who have recently participated in two research studies, co-ordinated by the LDC, who have consented to being contacted for future research studies that they may be eligible for. Our PPI committee has also recommended approaching at-risk groups, such as slimming clubs/weight watchers. Therefore we will contact such groups within the local community and the research team will run recruitment fares in those groups who agree.

   Additional awareness and interest in the study will be generated through locally organized events for Clinicians, GPs, nurses and other health care professionals. Further members of the research team will partake in other appropriate community events and meetings to publicise the study and distribute information. We will create a study website which will contain basic study information and a link to the most recent patient Information sheet, with a contact us button allowing patients to self-refer directly to the study team via email. We will also create a link to this study on the Leicestershire diabetes website that is designed and maintained by our group (http://www.leicestershirediabetes.org.uk), the NIHR Leicester Cardiovascular BRU and the NIHR Leicester-Loughborough Diet, Lifestyle and physical activity BRU. We will provide some background information about this area of research, what the study is about the inclusion criteria and contact details for further information. This will all be written in lay terminology as per usual for these websites. Previous studies conducted by our group have also had success by advertising the study on the UHL Trusts and the University of Leicester intra-net which we will also do for this study. This involves a small advertisement with the study logo, name very brief synopsis and contact details of the research team. Anyone interested can then request further information. They will be sent a postal invitation pack should they express interest and met the basic inclusion/exclusion criteria. We will recruit members of the public who self-refer and who meet the inclusion/exclusion criteria. We will put posters advertising the study in other community settings such as GP practices (who agree), diabetes clinics pharmacies, gyms and notices boards. We will also use digital and social media (such as facebook and twitter) to help promote the study, whilst interest and patient feedback regarding the study will be generated via other media outlets (e.g. press releases, radio) where possible.

   Healthy controls will be recruited through posters advertising the study in the University and the Trust, both of which have diverse ethnic staff groups, and through the study advertisements listed above.

ELIGIBILITY:
Inclusion Criteria:

* Capacity to provide informed consent before any trial-related activities
* Established T2DM (≥3months)
* HbA1c ≤ 9% if on triple therapy or ≤ 10% on diet & exercise or monotherapy or dual therapy
* Current glucose lowering therapy either mono, dual or triple of any combination of metformin, sulphonylurea, DPP-IV inhibitor, GLP-1 therapy or an SGLT2 +/- diet and exercise
* Poorly managed diet controlled diabetes (with HbA1c > 6.5% , not currently taking any glucose lowering therapy, meeting BMI inclusion range)
* Body mass index > 30Kg/m2 or > 27.5 Kg/m2 (South Asian),
* Diagnosis of T2DM before the age of 60 years of age
* Age ≥18 and ≤ 65 years

Exclusion Criteria:

* • Diabetes duration >12 years
* Currently taking more than three glucose lowering therapies
* Weight-loss of >5kg in the preceding 6 months
* Stage 4 or 5 chronic kidney disease (eGFR< 30ml/min/1.73m2),
* Current therapy with Insulin, thiazolidinediones, steroids or atypical antipsychotic medication
* Untreated thyroid disease
* Known macrovascular disease including coronary artery disease, stroke/TIA or peripheral vascular disease
* Presence of arrhythmia (including atrial fibrillation, atrial flutter, or 2nd or 3rd degree atrioventricular block)
* Known heart failure
* Other clinically relevant heart disease
* Inability to exercise or undertake a MRP
* Absolute contraindication to CMR
* Cardiovascular symptoms (angina, limiting dyspnoea during normal physical activity)
* Inflammatory condition e.g. Connective tissue disorder, Rheumatoid arthritis

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2015-10-02 (Actual); Primary Completion 2028-08-31 (Estimated); Study Completion 2028-08-31 (Estimated)

PRIMARY OUTCOMES:
Increase in circumferential PEDSR rate as measured by CMR at 12 weeks. | 12 weeks
  The aim of these analyses is to compare the primary outcome (diastolic strain rate) measured by CMR at 12 weeks between the TDR and standard care arms, and between the exercise and standard care arms. The primary analysis will be a per protocol analysis as this is a proof of principle study where we are primarily interested in the size of the treatment effect, rather than the practicability of the intervention.

SECONDARY OUTCOMES:
Left ventricular mass | Baseline, 4 and 12 weeks
  CMR to determine: structure and function
End diastolic volume | Baseline, 4 and 12 weeks
  CMR to determine: structure and function
End systolic volume | Baseline, 4 and 12 weeks
  CMR to determine: structure and function
Ejection Fraction | Baseline, 4 and 12 weeks
  CMR to determine: structure and function
LA Volumes | Baseline, 4 and 12 weeks
  CMR to determine: structure and function
Myocardial Systolic strain (Circumferential & Longitudinal) | Baseline, 4 and 12 weeks
  CMR to determine: structure and function
Systolic Strain Rates | Baseline, 4 and 12 weeks
  CMR to determine: structure and function
Mean Ascending & Descending Aortic Distensibility | Baseline, 4 and 12 weeks
  CMR to determine: arterial stiffness
Pulse-wave velocity | Baseline, 4 and 12 weeks
  CMR to determine: arterial stiffness
Global Myocardial Perfusion Reserve | Baseline, 4 and 12 weeks
  CMR to determine: structure and function, as a marker of vascular function
Myocardial triglyceride content | Baseline, 4 and 12 weeks
  CMR to determine: structure and function
Liver triglyceride content | Baseline, 4 and 12 weeks
  CMR to determine: structure and function
Extracellular volume (ECV) | Baseline, 4 and 12 weeks
  CMR to determine: structure and function, ECV as a marker of diffuse fibrosis
Mitral Inflow Velocity | Baseline, 4 and 12 weeks
  Echocardiography
Myocardial Relaxation | Baseline, 4 and 12 weeks
  Echocardiography
Non-Invasive Marker of Left Ventricular Filling Pressure | Baseline, 4 and 12 weeks
  Echocardiography
Abdominal Subcutaneous (Deep) distribution | 0 (consultation), 4 and 12 weeks
  MRI/CMR
Abdominal Subcutaneous (Superficial) distribution | 0 (consultation), 4 and 12 weeks
  MRI/CMR
Adiposity (Total Body Fat) | 0 (consultation), 4 and 12 weeks
  DEXA scan
Adiposity (Fat Free Mass) | 0 (consultation), 4 and 12 weeks
  DEXA scan
Physical Fitness & activity (Peak VO2max) | Baseline, 4 weeks and 12 weeks
  Cardiorespiratory fitness by incremental exercise testing (VO2max)
Physical Fitness & activity (Accelerometer) | Baseline, 4 weeks and 12 weeks
  Cardiorespiratory fitness by accelerometer for activity and sedentary time
Family & Full Medical History | Baseline
  diabetes diagnosis, duration, family history of CVD, diabetes type 1 & 2, stroke, myocardial infarction etc. Current medications.
HbA1c | Baseline, 4weeks, 12 weeks
  Biochemical Variables
Fasting Glucose | Baseline, 1 week, 2 week, 4weeks, 12 weeks
  Biochemical Variables
Insulin | Baseline, 4weeks, 12 weeks
  Biochemical Variables
Adiponectin | Baseline, 4weeks, 12 weeks
  Biochemical Variables
Leptin | Baseline, 4weeks, 12 weeks
  Biochemical Variables
Total Cholesterol | Baseline, 4weeks, 12 weeks
  Biochemical Variables
LDL (Low density lipoprotein) | Baseline, 4weeks, 12 weeks
  Biochemical Variables
HDL (High density lipoprotein) | Baseline, 4weeks, 12 weeks
  Biochemical Variables
Triglycerides | Baseline, 4weeks, 12 weeks
  Biochemical Variables
Liver Function Test (LFT) | Baseline, 4weeks, 12 weeks
  Biochemical Variables
Thyroid Function Tests (TFT) | Baseline, 4weeks, 12 weeks
  Biochemical Variables
Vitamin C | Baseline, 4weeks, 12 weeks
  Biochemical Variables
Vitamin D | Baseline, 4weeks, 12 weeks
  Biochemical Variables
Group B Vitamin Panel | Baseline, 4weeks, 12 weeks
  Biochemical Variables
Iron | Baseline, 4weeks, 12 weeks
  Biochemical Variables
Serum Ferritin | Baseline, 4weeks, 12 weeks
  Biochemical Variables
Full Blood Count (with Haematocrit) | Baseline, 4weeks, 12 weeks
  Biochemical Variables
B-Type Natriuretic Peptide (BNP) | Baseline, 4weeks, 12 weeks
  Biochemical Variables
Metabolomic and Inflammatory Markers | Baseline, 4weeks, 12 weeks
  Biochemical Variables
C-peptide | Baseline, 4weeks, 12 weeks
  Biochemical Variables
Height | Baseline
  Standard Anthropometric Variables
Weight | Baseline, 1, 2, 4, 6, 8, 12 weeks, 26 weeks, 52 weeks
  Standard Anthropometric Variables, derivation of BMI
Waist & Hip Circumference | Baseline, 12 weeks
  Standard Anthropometric Variables
Systolic and Diastolic BP | Baseline, 1, 2, 4, 6, 8, 12 weeks, 26 weeks, 52 weeks
  Standard Anthropometric Variables
Heart rate | Baseline, 1, 2, 4, 6, 8, 12 weeks, 26 weeks, 52 weeks
  Standard Anthropometric Variables
Hypoglycaemia | Baseline, 4weeks, 12 weeks
  self reported in blood glucose monitoring/hypo diary
7-Point Profile Glucose Monitoring | 0weeks, 4weeks, 12 weeks
  self reported in blood glucose monitoring/hypo diary
Adverse Events | Baseline, 1, 2, 4, 6, 8, 12 weeks
  Safety
Food Diary | Baseline, 12 weeks
  Self-reporting
EQ5D Questionnaire | Baseline, 12 weeks
  Questionnaire
Exercise Questionnaire | Baseline, 12 weeks
  Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Gerry Dr McCann, MD, Principal Investigator — University of Leicester
Locations (1):
- Glenfield Hospital (University Hospitals of Leicester NHS Trust), Leicester, United Kingdom

REFERENCES:
- [Result] Khan JN, Wilmot EG, Leggate M, Singh A, Yates T, Nimmo M, Khunti K, Horsfield MA, Biglands J, Clarysse P, Croisille P, Davies M, McCann GP. Subclinical diastolic dysfunction in young adults with Type 2 diabetes mellitus: a multiparametric contrast-enhanced cardiovascular magnetic resonance pilot study assessing potential mechanisms. Eur Heart J Cardiovasc Imaging. 2014 Nov;15(11):1263-9. doi: 10.1093/ehjci/jeu121. Epub 2014 Jun 26. PMID 24970723
- [Derived] Brady EM, Cao TH, Moss AJ, Athithan L, Ayton SL, Redman E, Argyridou S, Graham-Brown MPM, Maxwell CB, Jones DJL, Ng L, Yates T, Davies MJ, McCann GP, Gulsin GS. Circulating sphingolipids and relationship to cardiac remodelling before and following a low-energy diet in asymptomatic Type 2 Diabetes. BMC Cardiovasc Disord. 2024 Jan 3;24(1):25. doi: 10.1186/s12872-023-03623-y. PMID 38172712
- [Derived] Athithan L, Gulsin GS, Henson J, Althagafi L, Redman E, Argyridou S, Parke KS, Yeo J, Yates T, Khunti K, Davies MJ, McCann GP, Brady EM. Response to a low-energy meal replacement plan on glycometabolic profile and reverse cardiac remodelling in type 2 diabetes: a comparison between South Asians and White Europeans. Ther Adv Endocrinol Metab. 2023 Oct 6;14:20420188231193231. doi: 10.1177/20420188231193231. eCollection 2023. PMID 37811525
- [Derived] Alfuhied A, Gulsin GS, Athithan L, Brady EM, Parke K, Henson J, Redman E, Marsh AM, Yates T, Davies MJ, McCann GP, Singh A. The impact of lifestyle intervention on left atrial function in type 2 diabetes: results from the DIASTOLIC study. Int J Cardiovasc Imaging. 2022 Sep;38(9):2013-2023. doi: 10.1007/s10554-022-02578-z. Epub 2022 Mar 2. PMID 35233724
- [Derived] Walters GWM, Redman E, Gulsin GS, Henson J, Argyridou S, Yates T, Davies MJ, Parke K, McCann GP, Brady EM. Interrelationship between micronutrients and cardiovascular structure and function in type 2 diabetes. J Nutr Sci. 2021 Oct 4;10:e88. doi: 10.1017/jns.2021.82. eCollection 2021. PMID 34733500
- [Derived] Gulsin GS, Swarbrick DJ, Athithan L, Brady EM, Henson J, Baldry E, Argyridou S, Jaicim NB, Squire G, Walters Y, Marsh AM, McAdam J, Parke KS, Biglands JD, Yates T, Khunti K, Davies MJ, McCann GP. Effects of Low-Energy Diet or Exercise on Cardiovascular Function in Working-Age Adults With Type 2 Diabetes: A Prospective, Randomized, Open-Label, Blinded End Point Trial. Diabetes Care. 2020 Jun;43(6):1300-1310. doi: 10.2337/dc20-0129. Epub 2020 Mar 27. PMID 32220917
- [Derived] Gulsin GS, Brady EM, Swarbrick DJ, Athithan L, Henson J, Baldry E, McAdam J, Marsh AM, Parke KS, Wormleighton JV, Levelt E, Yates T, Bodicoat D, Khunti K, Davies MJ, McCann GP. Rationale, design and study protocol of the randomised controlled trial: Diabetes Interventional Assessment of Slimming or Training tO Lessen Inconspicuous Cardiovascular Dysfunction (the DIASTOLIC study). BMJ Open. 2019 Mar 30;9(3):e023207. doi: 10.1136/bmjopen-2018-023207. PMID 30928925
- [Derived] Gulsin GS, Swarbrick DJ, Hunt WH, Levelt E, Graham-Brown MPM, Parke KS, Wormleighton JV, Lai FY, Yates T, Wilmot EG, Webb DR, Davies MJ, McCann GP. Relation of Aortic Stiffness to Left Ventricular Remodeling in Younger Adults With Type 2 Diabetes. Diabetes. 2018 Jul;67(7):1395-1400. doi: 10.2337/db18-0112. Epub 2018 Apr 16. PMID 29661781
- See also: Leicester Diabetes Centre — http://www.leicestershirediabetes.org.uk